CLINICAL TRIAL: NCT03516318
Title: Using Social Media to Improve ART Retention and Treatment (SMART) Outcomes Among Youth Living With HIV (YLHIV) in Nigeria - The Youth SMART Study
Brief Title: Using Social Media to Improve ART Retention and Treatment Outcomes Among YLHIV in Nigeria
Acronym: Y-SMART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study funding ended before last round of data collection could be complete.
Sponsor: FHI 360 (Other)
Collaborators: Center for Population and Reproductive Health, University of Ibadan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1151489
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Youth; Social support; Social media; Retention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART Connections (Experimental): The intervention components include:
  * Informational messages that reflect the content of the structured group counseling curriculum and are posted to the Facebook group wall on a regular basis for approximately 4 to 5 months
  * Moderated, closed group chats in a "secret" Facebook group where YLHIV can interact with their peers and with a trained support group facilitator
  * Access to a trained facilitator via Facebook Messenger for the duration of the intervention who will be able to provide information or basic counseling on ART/HIV care related issues, with referral to health care services as needed
  Interventions: Behavioral: SMART Connections
- Control (No Intervention): All study participants, in both study arms, will receive standard services currently available to YLHIV in these facilities and communities. The services currently include: routine clinical care for HIV treatment including laboratory testing (CD4, viral load tests); active case management by community volunteers with intensive adherence support during the first 4 weeks of ART; adherence support through phone calls and SMS (short messaging service) reminders; and enhanced adherence counseling for patients with unsuppressed viral loads.

INTERVENTIONS:
Behavioral: SMART Connections — SMART Connections: Trained facilitators will deliver key informational messages and moderate online group discussions. The informational messages have been developed from key messages identified in each of the Positive Connections curriculum sessions. Each SMART Connections group will consist of approximately 15 to 20 YLHIV. Each online support group will begin with one in-person group meeting with the facilitator. During this meeting, participants meet one another and the facilitators. Facilitators will describe the intervention and set ground rules for participation. Ground rules will be discussed and accepted by the group members, but at a minimum, group members will be advised not to talk about what is discussed in the online group with people outside of the group.
  Arms: SMART Connections

SUMMARY:
A randomized control trial to test the effectiveness of a structured online support group, SMART (Social Media to improve ART Retention in Treatment) Connections, to improve retention in HIV care services among youth living with HIV (YLHIV) in Nigeria.

DETAILED DESCRIPTION:
Study aim is to examine the effect of an online structured support group intervention (SMART Connections) designed to improve retention in HIV care services among youth ages 15-21 years living with HIV enrolled in ART services. A randomized control trial in which youth living with HIV (YLHIV) will be allocated to standard of care (control) or standard of care plus an online support group and followed for 12 months. Structured questionnaires will be administered to participants at baseline, 6 and 12 months. Clinical data will also be extracted on participants. In-depth interviews with a subset of participants and intervention implementers will be completed at the end of the intervention period. Although participants will be recruited from health facilities, the intervention is conducted "virtually," by trained facilitators, not within the health facilities.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive and know their status
* Actively on ART for less than 12 months, including newly initiating patients
* Age 15 to 24 years
* Can demonstrate basic literacy necessary to participate in online chats

Exclusion Criteria:

* Unable to attend the initial intervention group meeting for treatment participants
* Currently enrolled in another research study related to HIV service retention or ART adherence
* Critically or severely ill requiring hospitalization or such that the individual is unable to provide informed consent at the time of study recruitment

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 355 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
12-month retention in HIV services | 12 months
  This main outcome is defined as the proportion of study participants retained in clinical HIV services and on treatment at 12 months after enrollment. We will abstract data from the clinic electronic medical record system on date of all visits, which are typically monthly, to ART services between enrollment and the end-line of this study.
  Retention is defined as having attended a scheduled HIV clinic visit within three months of the visit date. For our primary analysis, using a survival analysis approach, we will record the dates for all scheduled clinic visits for each participant, then follow the data up to three months from the date of the last visit attended. If a participant fails to return after a scheduled visit for more than three months, the date of the missed visit will be the date of loss to follow-up recorded, unless a death or transfer of service is documented.

SECONDARY OUTCOMES:
Social support score | 12 months
  To measure social support, we will use the Medical Outcomes Study - Social Support Survey (MOS-SSS).The MOS-SSS is a 19-item scale that covers the dimensions of emotional/informational (8 items), affectionate (3 items) and tangible (4 items) social support in addition to positive social interaction (3 items), and one additional item. Each item is measured on a 4 point Likert-type scale.From the scale a total SS score is calculated by summing the items. A transformed score can be calculated for total SS or each dimension by taking the raw score (total summed score), subtracting the number of items for the score and dividing by the total possible score for those items.
Adherence to antiretroviral treatment | 12 months
  Proportion of participants who are adherent to ART will be measured through self-reported measures in the structured questionnaire of treatment adherence and challenges with taking medication as prescribed. We will measure self-reported adherence using the AIDS Clinical Trials Group adherence measure (AACTG baseline: http://caps.ucsf.edu/uploads/tools/surveys/pdf/2098.4186.pdf). We will also extract viral load cell data from patient medical records to triangulate self-reported adherence. For this secondary outcome, a dichotomous variable will be created defined as adherent or not adherent (missed any doses of medication) in the prior 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Dulli, PhD, Principal Investigator — FHI 360 (Family Health International)
Locations (1):
- FHI 360, Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
De-identified, quantitative data on study participants will be uploaded to the USAID Development Data Library.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data on study participants will be shared once submission of the primary study manuscript has been completed, or no later than the end of project funding.
Access Criteria: Per the Development Data website: "Data submitted to the Development Data Library (DDL) will first be made available to USAID's (United States Agency for International Development) InfoGov Permanent Working Group (see ADS 579.2.d), the Operating Unit of Origin, and to clearance officials specified in ADS 579.3.2.5. Data sets that are determined (via the clearance process in ADS 579.3.2.5) to be "Public" are listed in the DDL, and the data itself and supporting documentation are made available to the global public. Data sets that are determined via the clearance process to be "Non-Public" or "Restricted Public" (see ADS 579.3.2.4) will be listed in the DDL only. Data sets tagged as Non-Public will remain unavailable to the public. Data sets tagged as Restricted will only be made available under certain use restrictions.
URL: http://www.usaid.gov/data

REFERENCES:
- [Derived] Dulli L, Ridgeway K, Packer C, Murray KR, Mumuni T, Plourde KF, Chen M, Olumide A, Ojengbede O, McCarraher DR. A Social Media-Based Support Group for Youth Living With HIV in Nigeria (SMART Connections): Randomized Controlled Trial. J Med Internet Res. 2020 Jun 2;22(6):e18343. doi: 10.2196/18343. PMID 32484444

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT03516318/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT03516318/SAP_001.pdf